CLINICAL TRIAL: NCT06917820
Title: Ultrasound-guided Clavipectoral Fascia Plane Block Versus Interscalene Brachial Plexus Block for Postoperative Analgesia in Midshaft Clavicular Surgery
Brief Title: Clavipectoral Block Versus Interscalene Block for Postoperative Analgesia in Midshaft Clavicular Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD142/2024
Record Dates: First submitted 2025-02-14; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Interscalene brachial plexus block group (Active Comparator): Peripheral nerve block Under sterile conditions, the high frequency probe will be positioned at the level of cricoid cartilage to visualize the brachial plexus between the anterior and middle scalene muscles. A total of 20 ml of local anesthetic (10 ml of bupivacaine 0.5% and 10 ml of normal saline) will be injected after negative aspiration, and needle will be adjusted to achieve its spread between the C5 and C6 nerve roots and between C6 and C7 nerve roots.
  Interventions: Procedure: Interscalene brachial plexus block
- Clavipectoral fascia plane block (Active Comparator): Peripheral nerve block Under sterile conditions, a high frequency linear probe will be initially placed over the anterior surface of the clavicle in a sagittal orientation. Essentially, there will be one injection on each side of the fracture after negative aspiration. The first injection will be 4-5 cm from the acromial end of the clavicle and the second one will be 4-5 cm from the sternal end of the clavicle. An in-plane technique will be used to view the needle advancing in a caudad to cephalad direction until it will rest on the clavipectoral fascia. The total amount of local anesthetic (LA) mixture will be 20 ml (10 ml of bupivacaine 0.5% and 10 ml of normal saline), divided into 10 ml medially and 10 ml laterally.
  Interventions: Procedure: Clavipectoral fascia plane block

INTERVENTIONS:
Procedure: Interscalene brachial plexus block — Ultrasound-guided peripheral nerve block that includes injection of local anesthetics between the C5 and C6 nerve roots and between C6 and C7 nerve roots.
  Arms: Interscalene brachial plexus block group
Procedure: Clavipectoral fascia plane block — Ultrasound-guided peripheral nerve block that includes injection of local anesthetics between the periosteum of clavicle and the surrounding clavipectoral fascia.
  Arms: Clavipectoral fascia plane block

SUMMARY:
The aim of this study is to compare between (ISBPB) and (CPB) as postoperative analgesic technique following midshaft clavicular fracture open reduction and internal fixation surgeries.

DETAILED DESCRIPTION:
The aim of this study is to compare between (ISBPB) and (CPB) as postoperative analgesic technique following midshaft clavicular fracture open reduction and internal fixation surgeries. Preoperative full precise medical history will be taken from patients. Routine investigations will be done to all patients including ECG and laboratory investigations as CBC, AST, ALT, INR, PT and PTT. Demographic data as age and weight will be recorded. All patients will be consented for every anesthetic and surgical procedure to be done. For all patients, on arrival to the operating room, ECG, heart rate (HR), non-invasive blood pressure, and pulse oximetry will be monitored. Patients will receive 0.03 mg/kg of IV midazolam as anxiolytic and 3 L/ min nasal oxygen.

Then, in supine position, the diaphragmatic excursion measurement will be performed on the hemidiaphragm at the same side of the study block. Excursion amplitude will be defined as the craniocaudal perpendicular distance from the minimum to the maximum point of diaphragm excursion. Diaphragmatic excursion measurements will be performed before induction of general anesthesia and performing the block technique and at 3 hours after the block or 1 hour after recovery from anesthesia if the surgery lasted more than 2 hours.

After that, induction of GA will be performed by injecting intravenous (IV) 1 mcg/kg fentanyl, 2 mg/kg propofol and 0.5 mg/kg atracurium.

Then, the patients will receive one of the study blocks as following:

Group A: This group will receive ultrasound-guided clavipectoral fascia plane block.

Group B: This group will receive ultrasound-guided interscalene plexus block.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged from 21 to 60 years.
* American Society of Anesthesiologists (ASA) class I and II status.
* Of both sexes.
* Patients undergoing elective midshaft clavicle fracture open reduction and internal fixation surgery.

Exclusion Criteria:

* Patient refusal.
* American Society of Anesthesiologists (ASA) class llI and IV status.
* Patients with bleeding disorders.
* A history of relevant drug allergy to any of the used drugs.
* Alcohol or drug abuse and opioid dependence.
* Pregnant female patients.
* Patients with BMI above 30 kg/m2.
* Patients with infection at site of the fracture or the block procedure.
* Patients with reduced pulmonary functions due to chronic obstructive pulmonary disease (COPD), uncontrolled asthma, pneumothorax or pleural effusion.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Time to first rescue analgesia | 24 hours after injection
  The time to first rescue analgesia with time frame of 24 hours after the study block will be recorded.
Rescue analgesia consumed | 24 hours after injection
  The total dose of rescue analgesia consumed within 24 hours after the block will be recorded.

SECONDARY OUTCOMES:
Incidence of hemi-diaphragmatic paralysis | 3 hours after block or 1 hour after recovery from anesthesia.
  The incidence of hemi-diaphragmatic paralysis at 3 hours after block or 1 hour after recovery from anesthesia if the surgery lasted more than 2 hours. Hemi-diaphragmatic paralysis will be defined as greater than 50% reduction in diaphragmatic excursion compared with the pre block value during deep breathing.
Visual analogue scale (VAS) | 24 hours after injection
  The VAS is psychometric measuring instrument designed to document the disease-related symptom severity in individual patients. It will be recorded at 4-hour intervals. A VAS score of 4 or more will be treated with pethidine 50 mg IM as rescue analgesia to be repeated if needed provided that the total 24-hour dosage will not exceed 150 mg.
Heart rate | 24 hours after injection
  The heart rate of patients will be recorded at baseline just after the block and at the same intervals as the VAS.
Mean arterial blood pressure | 24 hours after injection.
  The mean arterial blood pressure of patients will be recorded at baseline just after the block and at the same intervals as the VAS.
Motor function of the relevant upper limb | 3 hours after block or 1 hour after recovery from anesthesia.
  Motor function of the relevant upper limb will be evaluated before induction of general anesthesia and performing the block technique and at 3 hours after the block or 1 hour after recovery from anesthesia if the surgery lasted more than 2 hours in the distribution of the axillary nerve (shoulder abduction), musculocutaneous nerve (elbow flexion), radial nerve (wrist extension), median nerve (wrist flexion), and ulnar nerve (thumb/finger adduction) using a 3-point scale (0 = normal strength, 1 = paresis, or 2 = paralysis), with maximal total motor block score of 10.
Other complications | 24 hours after injection
  Complications like postoperative nausea and vomiting, Horner's syndrome and pneumothorax will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Moustafa K Reyad, Professor, Study Director — Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No